CLINICAL TRIAL: NCT04914663
Title: All-extremity Exercise as a Novel Strategy for Optimizing Cardiovascular Function During Chemotherapy for Breast Cancer
Brief Title: All-extremity Exercise During Breast Cancer Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB202100182 -N; 1R21HL152264-01A1 (NIH); PRO00031309 (Other: University of Florida); OCR40536 (Other: UF OnCore)
Record Dates: First submitted 2021-05-28; First posted 2021-06-04 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- All-extremity exercise (Experimental)
  Interventions: Behavioral: Exercise training
- Treadmill exercise (Active Comparator)
  Interventions: Behavioral: Exercise training
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Exercise training — Exercise training performed at home under remote live supervision over 12 weeks while patients undergo chemotherapy for breast cancer.
  Arms: All-extremity exercise; Treadmill exercise

SUMMARY:
Currently, there are 3.5 million breast cancer survivors in the United States and this number is expected to increase dramatically. The proposed research will examine whether a novel exercise intervention for breast cancer patients who are undergoing chemotherapy protects against cardiovascular dysfunction. Findings may have implications for cardiovascular disease prevention in this population.

ELIGIBILITY:
Inclusion Criteria:

* Active diagnosis of primary invasive non-metastatic breast cancer, stages I-III
* Female
* 18 to 85 years of age
* Scheduled to initiate neoadjuvant or adjuvant chemotherapy (anthracycline, alkylating agent and/or taxane)
* Absence of contraindications to exercise
* Study clinician approval
* Able to give consent
* Informed consent obtained from the subject and documentation of subject agreement to comply with study-related process

Exclusion Criteria:

* Do not meet inclusion criteria
* Receiving targeted therapies (CDK4/6 or PARP inhibitors)
* Receiving radiation therapy concurrent with chemotherapy
* Lymphedema stage ≥ 2 prior to study enrollment
* Any relevant cardiovascular diseases (stroke, heart failure, myocardial ischemia during maximal graded exercise test, myocardial infarction, angina pectoris, coronary artery bypass surgery or angioplasty or coronary stent)
* Current participation in other experimental interventions that may confound interpretation of study findings (e.g., dietary intervention for weight loss)

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who will receive chemotherapy for breast cancer
Enrollment: 68 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in brachial artery FMD | 12 weeks
  Flow mediated dilation (FMD) is an established non-invasive measure of endothelial function. Brachial artery FMD will be determined via ultrasonography in response to reactive hyperemia following 5-min forearm ischemia.
Change in global longitudinal strain | 12 weeks
  Global longitudinal strain is a marker of acute subclinical cardiotoxicity and is recommended for monitoring cancer patients at risk of cancer therapy-related cardiac dysfunction.
Feasibility, tolerability and safety of exercise training during breast cancer chemotherapy | Monitored throughout the 12 weeks of intervention
  To evaluate the feasibility, tolerability and safety of all-extremity exercise compared with treadmill exercise in breast cancer patients undergoing chemotherapy, we will collect comprehensive information throughout the exercise intervention: completed vs. planned exercise dose (intensity/session, min/session, sessions/week), reasons for missed/partially completed sessions or study withdrawal, adverse events, and disease- and treatment-related outcomes. To specifically evaluate safety, should an adverse event occur, plans are in place for determination and monitoring according to the most recent National Cancer Institute Common Terminology Criteria for Adverse Events. Classification for seriousness, expectedness, severity and relationship to study intervention will be based on the NIH provided definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Demetra Christou, PhD, Principal Investigator — University of Florida
Locations (1):
- Integrative Cardiovasculal Physiology Laboratory, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No